CLINICAL TRIAL: NCT04023032
Title: Efficacy of a Multicomponent Cognitive Intervention Program on the Cognitive and Daily Function in Adults With Subjective Cognitive Decline and Mild Cognitive Impairments: A Pilot Study
Brief Title: Efficacy of a Multicomponent Cognitive Intervention in Adults With Subjective Cognitive Decline and Mild Cognitive Impairments
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 201805012RINA
Record Dates: First submitted 2019-07-15; First posted 2019-07-17 (Actual); Last update posted 2021-09-01 (Actual); Status verified 2021-01

CONDITIONS: Mild Cognitive Impairment; Subjective Cognitive Decline
MeSH Terms: conditions — Cognitive Dysfunction

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- multicomponent cognitive intervention (Experimental)
  Interventions: Behavioral: multicomponent cognitive intervention

INTERVENTIONS:
Behavioral: multicomponent cognitive intervention — The intervention takes place in groups of 6-10 participants and is leaded by one occupational therapist. It includes 16 sessions, 90 minutes each.
  The first part of each session starts with a 15-minute review of previous homework or relaxation. The second part, which lasts 35 minutes, involves structured training with activity-sheets, board games, role-playing and computerized games. The third part, which lasts 30 minutes, is the lifestyle interventions. The instructor explains the generalization of the previous activities toward daily life, and introduces healthy lifestyles. Through group discussions, the therapist guides participants to develop solutions and strategies for their memory or cognition-related problems and application to daily life. The last 10 minutes are used to suggest homework.

SUMMARY:
Individuals with mild cognitive impairment (MCI) and subjective cognitive decline (SCD) have greater risk of developing dementia. Cognitive intervention is a topic of great interest in individuals with MCI and SCD for the purpose of preventing or delaying the occurrence of dementia. There are many different types of cognitive interventions, which aim to positively impact the cognitive functioning of an individual and have been classified as cognitive stimulation, cognitive training, and cognitive rehabilitation. However, most studies used neuropsychological cognitive measures for outcome evaluation. The impact of cognitive interventions on daily functional performance among individuals with MCI and SCD were rarely explored. In addition, cognitive training focusing on specific cognitive outcomes is suspected to have limited far transfer to everyday measures. Therefore, a multicomponent intervention which integrates several types of intervention is recommended to reach the maximum impact on daily function.

The purposes of this study are to examine the effects of a multicomponent cognitive intervention on cognitive and daily functional outcomes in individuals with MCI and SCD, and to compare the effects between the two groups. In addition, the investigators will also investigate whether the demographic (e.g., age and educational level, etc.) and clinical variables (e.g., duration of cognitive complains, level of depression and baseline cognitive function, etc.) may affect the outcomes of cognitive intervention.

DETAILED DESCRIPTION:
This study is a pretest-posttest design. Thirty-five subjects with MCI and 35 with SCD, who are diagnosed by physicians, will be recruited from the neurology outpatient clinic of National Taiwan University Hospital. All participants will wait for 16 weeks as a historical control and then receive the multicomponent cognitive intervention. The intervention is composed of 14 weekly 1.5-hour group sessions and 2 individual sessions in a 4-month period.

The multicomponent cognitive intervention in this study is a combination of several approaches, including cognitive training, cognitive rehabilitation, lifestyle interventions, and psychological interventions. Cognitive training is an approach which trains patients by repeated practicing to optimize or restore cognitive functions. Cognitive rehabilitation is tailored programs in which therapist usually provides patient strategies focusing on specific activities of daily life. Lifestyle interventions educate and encourage individuals to make changes to their life to balance the risk and protective factors. The strategies can include regular physical exercise, healthy nutrition (i.e., Mediterranean diet), frequent participation in cognitively-stimulating activities, and reduction of smoking and heavy alcohol consumption. Psychological interventions target neuropsychiatric symptoms that are common among individuals with SCD and MCI (e.g., depression, anxiety, fatigue, poor sleep) and thus include relaxation exercises, mindfulness techniques, skills to manage stress and poor sleep, and cognitive behavioral techniques. By using the approaches above together, the investigators hope to improve participants' cognitive and daily function.

All participants will be assessed at four time points: before waiting period (A0), before the intervention (A1), right after the 16-week intervention (A2), and 16 weeks after the intervention (A3). The primary outcomes are the subjective and objective performance of activities of daily living, and the secondary outcomes are the cognitive performance on the neurological tests, anxiety, and depression.

ELIGIBILITY:
Inclusion Criteria:

* over 50 years old
* years of education > 6
* mild cognitive impairment or subjective cognitive decline diagnosed by physician
* the Barthel Index scored 100
* the Montreal Cognitive Assessment (MoCA) > 18
* the UPSA-Brief > 50

Exclusion Criteria:

* without concurrent major or significant psychiatric disorders
* severe physical diseases which might affect cognitive functions
* difficult to follow instructions due to visual or hearing impairments

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2019-01-02 (Actual); Primary Completion 2021-08-29 (Actual); Study Completion 2021-08-29 (Actual)

PRIMARY OUTCOMES:
Change from Baseline the Brief University of California San Diego (UCSD) Performance-Based Skills Assessment (UPSA-Brief ) (Traditional Chinese Version) at 16 weeks, 32 weeks, and 48 weeks | baseline, 16th, 32nd and 48th week
  The UPSA-Brief, which consists of 2 subscales (communication and financial), is a useful performance-based functional outcome scale. It has adequate psychometric properties, predicts residential independence, is sensitive to change, and requires only 10-15 minutes to administer.
Change from Baseline the Activities of Daily Living Questionnaire at 16 weeks, 32 weeks, and 48 weeks | baseline, 16th, 32nd and 48th week
  The Activities of Daily Living Questionnaire (ADLQ) is an informant-based assessment of functional abilities in patients with probable Alzheimer disease and other forms of dementia. The ADLQ measures functioning in six areas: self-care, household care, employment and recreation, shopping and money, travel, and communication.
Change from Baseline the Contextual Memory Test (CMT) at 16 weeks, 32 weeks, and 48 weeks | baseline, 16th, 32nd and 48th week
  The CMT is used to objectively measure awareness of memory capacity, strategy use and recall in adults with memory dysfunction. It assess 3 areas of memory including: awareness of memory capacity, recall of line-drawn items, and strategy use.
Change from Baseline the Miami Prospective Memory Test (MPMT) at 16 weeks, 32 weeks, and 48 weeks | baseline, 16th, 32nd and 48th week
  The Miami Prospective Memory Test evaluates time-related and event-related prospective memory ability of older adults.
Change from Baseline the Everyday Memory Questionnaire (EMQ) at 16 weeks, 32 weeks, and 48 weeks | baseline, 16th, 32nd and 48th week
  The Everyday Memory Questionnaire (EMQ) was developed as a subjective measure of memory failure in everyday life.
Change from Baseline the Cognitive Failure Questionnaire (CFQ) at 16 weeks, 32 weeks, and 48 weeks | baseline, 16th, 32nd and 48th week
  The CFQ assesses the frequency with which people experienced cognitive failures in daily life.

SECONDARY OUTCOMES:
Change from Baseline the Word Sequence Learning Test at 16 weeks, 32 weeks, and 48 weeks | baseline, 16th, 32nd and 48th week
Change from Baseline the Wechsler Memory Scale-3rd ed. (WMS-III) Logical Memory (LM) subtest at 16 weeks, 32 weeks, and 48 weeks | baseline, 16th, 32nd and 48th week
Change from Baseline the Wechsler Memory Scale-3rd ed. (WMS-III) Family Pictures (FP) subtest at 16 weeks, 32 weeks, and 48 weeks | baseline, 16th, 32nd and 48th week
Change from Baseline the Color Trails Test at 16 weeks, 32 weeks, and 48 weeks | baseline, 16th, 32nd and 48th week
Change from Baseline the Geriatric Depression Scale-Short Form (GDS-S) at 16 weeks, 32 weeks, and 48 weeks | baseline, 16th, 32nd and 48th week
Change from Baseline the State-Trait Anxiety Inventory-Situation (STAI-S) at 16 weeks, 32 weeks, and 48 weeks | baseline, 16th, 32nd and 48th week

CONTACTS AND LOCATIONS:
Overall Officials: Hui-Fen Mao, Principal Investigator — National Taiwan University Hospital
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No